CLINICAL TRIAL: NCT02068547
Title: Bone Marrow Aspirate Concentration in Posterior Cervical Fusion
Acronym: BMAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor closed study due to low enrollment
  Sponsor closed study due to low enrollment
  Sponsor closed study due to low enrollment.
Sponsor: Washington University School of Medicine (Other)
Collaborators: Harvest Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201308043
Record Dates: First submitted 2014-02-17; First posted 2014-02-21 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Cervical Myelopathy; Radiculopathy
Keywords: posterior cervical fusion; posterior cervical decompression
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - Surigical Best Practice (Active Comparator): Group 1 will receive current best practice for posterior instrumented fusion (locally harvested autograft, demineralized bone matrix, and cadaveric allograft)
  Interventions: Biological: locally harvested autograft, demineralized bone matrix, and cadaveric allograft
- Group 2 - autograft/BMAC (Experimental): Group II, will receive locally harvested autograft and 20 cc of bone marrow aspirate concentration.
  Interventions: Biological: Bone Marrow Aspirate

INTERVENTIONS:
Biological: locally harvested autograft, demineralized bone matrix, and cadaveric allograft
  Arms: Group 1 - Surigical Best Practice
Biological: Bone Marrow Aspirate
  Arms: Group 2 - autograft/BMAC

SUMMARY:
The purpose of this research is to test if that combining bone marrow aspirate (removing bone marrow with a needle) concentration with locally harvested (collected) autograft (patient's own bone from another part of the body) for use as the bone graft results in equal rates of a successful procedure (fusion), as compared to current best practice in high-risk patients undergoing posterior cervical fusion.

Hypothesis: Bone marrow aspirate concentration combined with locally harvested autograft results in equivalent rates of bony fusion, as compared to current best practice in high-risk patients undergoing posterior cervical decompression and fusion.

DETAILED DESCRIPTION:
100 consecutive high-risk patients who meet the following inclusion criteria: are 18-75 years of age, require a cervical spine MRI as part of their standard of care show evidence of CSM, and have cervical alignment allowing posterior instrumented fusion. High-risk will be defined as having a diagnosis of rheumatoid arthritis, osteoporosis, current smoker, or BMI >30. Patients will be excluded if they have any MRI incompatible devices, have any prior cervical instrumentation, require an instrumented anterior cervical fusion, or have an underlying neurological condition affecting the cervical spine (MS, ALS, HIV).

Patients will be sequentially randomized to one of two treatment groups. Group I, will receive current best practice for posterior instrumented fusion (locally harvested autograft, demineralized bone matrix, and cadaveric allograft). Group II, will receive locally harvested autograft and 20 cc of bone marrow aspirate concentration. To assist with analysis, we will collect information from patients' hematology results, obtained per their standard of care pre-operative workup. All patients will be treated post-operatively at the discretion of the treating surgeon. All patients will follow-up at 6 weeks, 3 months, 6 months, 12 months, and 24 months. At the 6, 12, and 24-month follow-up all patients will undergo flexion/extension X-rays, fusion will be defined as less than 2 mm or motion. A cervical spine CT may also be obtained at 24 months on all patients to assess fusion at the discretion of the treating surgeon. All radiographic assessments of fusion will be made by a Washington University staff radiologist, blinded to patient treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75
* Have at least one of the following high risk qualifications: BMI >30, Rheumatoid Arthritis, Osteoporosis, Current smoker
* Able to cooperate in the completion of standardized outcome measures (multiple questionnaires)
* Willing and able to comply with study protocol
* Symptomatic cervical myelopathy and/or radiculopathy
* Scheduled for cervical alignment, allowing management with a posterior approach

Exclusion Criteria:

* MRI incompatible device
* History of prior cervical instrumentation
* Requires an instrumented anterior cervical fusion
* History of underlying neurological condition affecting the cervical spine (MS, Amyotrophic Lateral Sclerosis, HIV)
* Pre-existent neurologic disorder or mental disorder that would preclude accurate evaluation (psychiatric disease, Parkinson's disease, Alzheimer's disease)
* History of previous cervical fusion at the operative site
* Pregnant
* Active malignancy
* Previous history of posterior cervical decompression

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Z Ray, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Washington University in St. Louis School of Medicine, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Groups:
- Autograft/DBM/Cadaver Allo: Group 1 will receive current best practice for posterior instrumented fusion (locally harvested autograft, demineralized bone matrix, and cadaveric allograft)
  locally harvested autograft, demineralized bone matrix, and cadaveric allograft
- Autograft/BMAC: Group II, will receive locally harvested autograft and 20 cc of bone marrow aspirate concentration.
  Bone Marrow Aspirate
Period: Overall Study
Arm/Group | Autograft/DBM/Cadaver Allo | Autograft/BMAC
Started | 4 | 4
Completed | 0 | 1
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 3 | 3
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Surigical Best Practice: Group 1 will receive current best practice for posterior instrumented fusion (locally harvested autograft, demineralized bone matrix, and cadaveric allograft)
  locally harvested autograft, demineralized bone matrix, and cadaveric allograft
- Group 2: Group II, will receive locally harvested autograft and 20 cc of bone marrow aspirate concentration.
  Bone Marrow Aspirate
- Total: Total of all reporting groups
Arm/Group | Surigical Best Practice | Group 2 | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 53.09 [36.84 to 67.33] | 59.75 [55.87 to 62.66] | 56.42 [36.84 to 67.33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Rate of Fusion
Description: Rate of fusion - (6, 12, and 24 months) Rate of fusion will be assessed by flexion extension X-rays at routine follow-up, translation method (<2mm) and/or by computed tomography (CT) scan at 2 year post-operatively.
Time Frame: 6 months, 12 months, 24 months
Population: Study was discontinued prior to data being analyzed.
Arm/Group | Surigical Best Practice | Group 2
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Physical and Mental Health From Subject's Point of View
Description: Short Form 36 (SF-36) is a profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index.
Time Frame: 24 months
Population: Study was discontinued prior to data being analyzed.
Arm/Group | Surigical Best Practice | Group 2
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Neck Pain Affects Every Day Activities
Description: Questionnaire that helps determine how a subject's neck pain affects their ability to manage every day activities.
Time Frame: 24 Months
Population: Study was discontinued prior to data being analyzed.
Arm/Group | Surigical Best Practice | Group 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: There were no adverse events to report.
Arm/Group | Surigical Best Practice | Group 2
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT02068547/Prot_SAP_000.pdf